CLINICAL TRIAL: NCT03133975
Title: Vitamin D Supplementation for Reduction of Dyslipidemia in Premenopausal Women
Brief Title: Vitamin D Supplementation for Treatment of Dyslipidemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Eman Khashaba, Lecturer in Industrial Medicine, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R/17.03.86
Record Dates: First submitted 2017-04-26; First posted 2017-04-28 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Dyslipidemias
Keywords: high dose vitamin D; dyslipidemia; premenopausal women
MeSH Terms: conditions — Dyslipidemias | interventions — Cholecalciferol; Therapeutics; Proteins

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial VITAMIN D for treatment of dyslipedemia
Who Masked: Participant, Investigator
Masking Description: double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Single high dose IM VIT D
  Interventions: Drug: Vitamin D3 (Treatment)
- Control (Active Comparator): Usual diet mix of carbohydrates - lipid - protein - minerals & vitamins
  Interventions: Other: Mixed diet of carbohydrate and protein (Control)

INTERVENTIONS:
Drug: Vitamin D3 (Treatment) — Single high dose vitamin D3 in treatment of dyslipedemia
  Other Names: divarol
  Arms: Treatment
Other: Mixed diet of carbohydrate and protein (Control) — Mixed diet of carbohydrate and protein
  Arms: Control

SUMMARY:
This study will be conducted to Assess possible reduction in lipid profile (LDL-Triglecerides-cholesterol) among pre-menopausal women in vit D group compared to standard treatment group after 3 months & 6 month of follow up as prophylaxis step for atherosclerosis.

DETAILED DESCRIPTION:
Vitamin D receptor gene mutations have been associated with increased incidence of arterial hypertension. While, hyperlipidemia and lipoprotein oxidation in bone is leading to osteoporosis by inhibiting osteoblastic differentiation It has been reported that vitamin D supplementation has shown pro-atherogenic effects in rats, and its deficiency is associated with the deterioration of atherogenesis These contradictory findings on the progression of atherosclerosis were examined in this study.

Aim: This study will be conducted to assess possible reduction in lipid profile (LDL-Triglycerides-cholesterol) among pre-menopausal women in vitamin D group compared to standard treatment group after 3 months & 6 month of follow up as prophylaxis step for atherosclerosis.

Subject and methods: Randomized clinical trial with double blinding will be performed on two groups study group and control group. The cases will recruited from outpatient clinic of medicine department in Mansoura university Hospital.

Sample size: based on pilot study after start of trial

Study groups:

Intervention group: High dose vitamin D3 IM treatment group according to vitamin D3 level after laboratory assessment.

Standard treatment group: Balanced diet mix of Carbohydrate, lipid, protein and fat diet minerals and vitamins for same period of follow up.

Inclusion criteria : pre-menopausal females (35-45 years old)

* No co morbidity
* Negative history of contraceptive pills or drug history of cholesterol lowering drugs
* Absent chronic diseases

There is possible recruiting of postmenopausal women according to difficulty in finding pre-menopausal women.

Methods: study patients will be subjected to:

* Full history taking,clinical examination, Anthropometric measurements.
* Laboratory investigations: Vitamin D3 assessment for all study patients.

Outcome that will be measured before and after follow up:

1. Serum 25 hydroxy Vitamin D3
2. C reactive protein
3. Serum Calcium level
4. Complete Lipid profile: LDL-HDL-Triglycerides -Total cholesterol quantitative and qualitative assessment.Patient will be fasting for at least 12-14 h then 5 mL venous blood sample will be drawn from each patient into plain tube and left to clot. Serum for routine analysis and the other aliquot will be stored at -21°C analysis will be separated by centrifugation into two aliquots; one will be used

ELIGIBILITY:
Inclusion Criteria:

* premenopausal females (35-45 years)

Exclusion Criteria:

* no co morbodity
* no lipid lowering drugs or contraceptive pills

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — to highlight the effect on females as it is more common among premenopausal women
Enrollment: 30 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
serum levels of LDL-HDL-Total cholesterol-triglecerides | 3 months-6 months
  reduction in lipid profile significantly than controls

CONTACTS AND LOCATIONS:
Overall Officials: Nibal Murad, lectURER, Principal Investigator — Mansoura University-Faculty of Medicine
Locations (1):
- Faculty of Medicine, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No